CLINICAL TRIAL: NCT02158520
Title: Randomized Phase II Study of AB (Nab-Paclitaxel [Abraxane?], Bevacizumab) Versus Ipilimumab for Therapy of Unresectable Stage IV Metastatic Malignant Melanoma
Brief Title: Nab-Paclitaxel and Bevacizumab or Ipilimumab as First-Line Therapy in Treating Patients With Stage IV Melanoma That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ACCRU RU261206I; NCI-2013-01112 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ML28605; RU261206I; ACCRU RU261206I (Other: Academic and Community Cancer Research United); P30CA015083 (NIH); NCT01879306 (obsolete NCT alias)
Record Dates: First submitted 2014-06-05; First posted 2014-06-09 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2019-02

CONDITIONS: Metastatic Melanoma; Mucosal Melanoma; Stage IV Cutaneous Melanoma AJCC v6 and v7; Stage IV Uveal Melanoma AJCC v7; Unresectable Melanoma
MeSH Terms: conditions — Melanoma; Uveal Melanoma | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Ipilimumab; CTLA-4 Antigen; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (bevacizumab and nab-paclitaxel) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and nab-paclitaxel IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients experiencing progressive disease may cross-over to Arm B within 2-4 weeks.
  Interventions: Biological: Bevacizumab; Other: Laboratory Biomarker Analysis; Drug: Nab-paclitaxel; Other: Pharmacological Study
- Arm B (ipilimumab) (Experimental): Patients receive ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients experiencing progressive disease may cross-over to Arm A within 2-4 weeks.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar QL 1101; BEVACIZUMAB, LICENSE HOLDER UNSPECIFIED; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
  Arms: Arm A (bevacizumab and nab-paclitaxel)
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
  Arms: Arm B (ipilimumab)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; paclitaxel albumin-stabilized nanoparticle formulation; Protein-bound Paclitaxel
  Arms: Arm A (bevacizumab and nab-paclitaxel)
Other: Pharmacological Study — Correlative studies

SUMMARY:
This randomized phase II trial studies how well nab-paclitaxel and bevacizumab or ipilimumab works as first-line therapy in treating patients with stage IV melanoma that cannot be removed by surgery. Drugs used in chemotherapy, such as nab-paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Bevacizumab may stop the growth of tumor cells by binding to a protein called vascular endothelial growth factor (VEGF) and by preventing the growth of new blood vessels that tumors need to grow. Ipilimumab blocks a substance called cytotoxic T-lymphocyte-associated antigen-4 (CTLA4) on the surface of T cells and may help the immune system kill cancer cells. It is not yet known whether nab-paclitaxel and bevacizumab is more effective than ipilimumab in treating melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess whether the combination nab-paclitaxel and bevacizumab (AB) prolongs progression-free status relative to ipilimumab as a treatment in patients with unresectable stage IV melanoma.

SECONDARY OBJECTIVES:

I. To estimate the hazard of death among those randomized to AB then ipilimumab relative to those randomized to ipilimumab then AB as treatment in patients with unresectable stage IV melanoma.

II. To assess whether tumor response rate (as determined by Response Evaluation Criteria in Solid Tumors [RECIST] criteria 1.1) differs with respect to first (1st) treatment course.

III. To estimate whether the tumor response rate differs with respect to second (2nd) treatment course for those who progressed during their first treatment course.

IV. To further examine the safety profile of each of these regimens.

CORRELATIVE OBJECTIVES:

I. To examine the pharmacokinetics of nab-paclitaxel when combined with bevacizumab therapy.

II. To examine pharmacodynamic changes of blood-derived parameters (biomarkers) of angiogenesis and immunity as a function of therapy.

III. To examine whether changes in serum biomarkers are also seen in the tumor.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive bevacizumab intravenously (IV) over 30-90 minutes on days 1 and 15 and nab-paclitaxel IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients experiencing progressive disease may cross-over to Arm B within 2-4 weeks.

ARM B: Patients receive ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients experiencing progressive disease may cross-over to Arm A within 2-4 weeks.

After completion of study treatment, patients are followed up for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic proof of surgically unresectable stage IV malignant melanoma - including that of uveal and mucosal origin

  * Note: biopsy can be of locoregional disease in setting of clinically evident stage IV disease; a biopsy of the primary tumor alone does not fulfill this requirement
* No more than 2 prior courses of systemic therapy for metastatic melanoma
* For patients with metastatic melanoma not of uveal origin, v-raf murine sarcoma viral oncogene homolog B1 (BRAF) V600 mutation determination using a Clinical Laboratory Improvement Amendments (CLIA)-approved testing method on metastatic tumor tissue

  * NOTE: patients with metastatic melanoma of uveal origin do not need to have formal BRAF testing due to low probability of a BRAF V600 mutation in their metastatic tumor
* Measurable disease; note: disease that is measurable by physical examination only is not eligible
* Life expectancy of >= 4 months
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Absolute neutrophil count >=1500/mL (obtained =< 14 days prior to registration/randomization)
* Platelet count >= 100,000 x 10^9/L (obtained =< 14 days prior to registration/randomization)
* Hemoglobin >= 9 g/dL (obtained =< 14 days prior to registration/randomization) (patients may be transfused to meet this requirement)
* Creatinine =< 1.5 x upper limit of normal (ULN) (obtained =< 14 days prior to registration/randomization); institutional norms are acceptable
* Total bilirubin =< 1.5 mg/dL (obtained =< 14 days prior to registration/randomization) (exception: patients with documented Gilbert?s syndrome are allowed to participate despite elevated bilirubin)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 2.5 x ULN and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2.5 x ULN (obtained =< 14 days prior to registration/randomization)
* Alkaline phosphatase =< 2.5 x ULN (obtained =< 14 days prior to registration/randomization); if bone metastasis is present in the absence of liver metastasis then =< 5 x ULN
* Urine dipstick for proteinuria < 2+ (obtained =< 14 days prior to registration/randomization) (patients discovered to have >= 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate =< 1 g of protein in 24 hours to be eligible)
* Negative serum pregnancy test done =< 7 days prior to registration/randomization, for women of childbearing potential only

  * Note:

    * Females: adequate contraception must be used by both patient and partner while receiving study drug and for 12 weeks after the last dose of study drug
    * Males: adequate contraception must be used by both patient and partner while receiving study drug; men who have a partner of childbearing age should also avoid fathering a child for 6 months after the last dose of study drug
* Ability to understand and the willingness to sign a written informed consent document
* Mayo Rochester patients only: willingness to provide mandatory blood samples for research purposes

Exclusion Criteria:

* Brain metastases per magnetic resonance imaging (MRI) or computed tomography (CT)

  * Note: patients who have had therapy for brain metastasis (i.e., surgical resection, whole brain radiation, or stereotactic radiosurgery [SRS] even if stable) are not eligible
* Other investigational agents =< 4 weeks prior to registration/ randomization
* Anti-cancer therapy (including immunotherapy) =< 4 weeks prior to registration/randomization; exception: adjuvant Leukine =< 14 days prior to registration/randomization
* Prior treatment in the adjuvant or metastatic setting with any of the following:

  * Agents disrupting VEGF activity or targeting vascular endothelial growth factor receptor (VEGFR);
  * Ipilimumab;
  * Or taxane based chemotherapy regimens (including paclitaxel, docetaxel, cabazitaxel or nab-paclitaxel)
* Major surgical procedure, open biopsy, or significant traumatic injury =< 4 weeks prior to registration/randomization; (port-a-cath placement does not count as a major surgical procedure and patients can be enrolled at any time after placement)
* Fine needle aspirations or core biopsies =< 7 days prior to registration/ randomization
* Planned/or anticipated major surgical procedure during the course of the study
* Other medical conditions including but not limited to:

  * History of liver disease such as cirrhosis, chronic active hepatitis, chronic persistent hepatitis or hepatitis B or C
  * Active infection requiring parenteral antibiotics
  * Poorly controlled high blood pressure (>= 150 mmHg systolic and/or 100 mmHg diastolic) despite treatment
  * New York Heart Association class II-IV congestive heart failure
  * Serious cardiac arrhythmia requiring medication
  * Myocardial infarction or unstable angina =< 6 months prior to registration/randomization
  * Clinically significant peripheral vascular disease
  * Deep venous thrombosis or pulmonary embolus =< 1 year of registration/randomization
  * Ongoing need for full-dose oral or parenteral anticoagulation
  * Ongoing anti-platelet treatment other than low-dose aspirin (i.e., aspirin 81 mg by mouth daily)
  * Active bleeding or pathological conditions that carry high risk of bleeding (e.g., known esophageal varices, etc.)
  * Serious, non-healing wound (including wounds healing by secondary intention), ulcer or bone fracture
  * History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess =< 6 months prior to registration/randomization
  * History of central nervous system (CNS) disease (e.g., vascular abnormalities, etc.), clinically significant stroke or transient ischemic attack (TIA) =< 6 months prior to registration/randomization, seizures not controlled with standard medical therapy
  * Radiographically documented tumor invading major blood vessels
  * History of hypertensive crisis or hypertensive encephalopathy
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men and women of reproductive potential who are not using effective birth control methods Note: women of childbearing potential must have a negative serum pregnancy test =< 7 days prior to registration/randomization; adequate contraception must be used while receiving study drug and for 12 weeks after the last dose of study drug, by both women and men and by both patient and partner; men who have a partner of childbearing potential should also avoid fathering a child for 6 months after the last dose of study drug
* Existence of peripheral sensory neuropathy >= grade 2 (from any cause)
* History of other malignancy =< 5 years with the exception of basal cell or squamous cell carcinoma of the skin, treated with local resection only, or carcinoma in situ (e.g. of the cervix, breast, prostate, etc.)
* Radiation therapy (other than palliative) =< 2 weeks prior to randomization; note: patients who have had > 25% of their functional bone marrow irradiated are not eligible for this trial
* Active or recent history of hemoptysis (>= 1/2 teaspoon of bright red blood per episode) =< 30 days prior to registration/randomization
* Known hypersensitivity to any of the components of ipilimumab, bevacizumab, or nab-paclitaxel
* History of inflammatory bowel disease (e.g., Crohn?s, ulcerative colitis) - note patients with irritable bowel syndrome are eligible
* Diagnosis of autoimmune disease (i.e., rheumatoid arthritis, scleroderma, systemic lupus erythematosus [SLE], autoimmune vasculitis, Guillain-Barre syndrome, etc.), regardless if patient is currently receiving treatment at time of registration/randomization
* Systemic corticosteroids use =< 2 weeks, regardless of indication; note: patients who are on inhaled corticosteroids are eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10-18 (Actual); Primary Completion 2017-05-24 (Actual); Study Completion 2019-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Svetomir N Markovic, Principal Investigator — Academic and Community Cancer Research United
Locations (13):
- United States (13):
  - Saint Mary's Medical Center, San Francisco, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Illinois, Chicago, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was closed to enroll on November 19, 2015 after having enrolled 24 patients (12 patients per arm) due to the FDA approval of new agents for this patient population.
Groups:
- Arm A (Bevacizumab and Nab-paclitaxel): Patients receive bevacizumab 10mg/kg IV over 30-90 minutes on days 1 and 15 and nab-paclitaxel 150 mg/m^2 IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients experiencing progressive disease may cross-over to Arm B within 2-4 weeks.
- Arm B (Ipilimumab): Patients receive ipilimumab 3 mg/kg IV over 90 minutes on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients experiencing progressive disease may cross-over to Arm A within 2-4 weeks.
Period: Overall Study
Arm/Group | Arm A (Bevacizumab and Nab-paclitaxel) | Arm B (Ipilimumab)
Started | 12 | 12
AE Evaluated Prior to Crossover | 12 | 12
Eligible for Crossover (Discontinued initial treatment due to disease progression) | 8 | 8
Eligible for Crossover With AE Evaluated (Patients eligible for crossover AND evaluated for adverse events) | 7 | 7
Crossover Cohort (Patients who experienced progressive disease and did crossover) | 4 | 6
Completed (Eligible patients) | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Bevacizumab and Nab-paclitaxel) | Arm B (Ipilimumab) | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Median (Full Range); unit: years] | 60 [37 to 77] | 61 [38 to 81] | 61 [37 to 81]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender: Male | 8 | 7 | 15
  Sex/Gender: Female | 4 | 4 | 8
  Sex/Gender: Unknown | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Prior radiation therapy [Count of Participants; unit: Participants] — Patients who received radiation therapy prior to study treatment
  Participants | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression free survival (PFS) is defined as the time from the date of randomization to the date of disease progression or death resulting from any cause, whichever comes first. Progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From randomization to the earliest documentation of progression as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria (version 1.1) or death from any cause without the documentation of progression, assessed up to 4 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm A (Bevacizumab and Nab-paclitaxel) | Arm B (Ipilimumab)
Number analyzed (Participants) | 12 | 12
days | 139 [86 to NA] — The 95% confidence interval upper limit was not reached (below the level of detection). | 94 [74 to NA] — The 95% confidence interval upper limit was not reached (below the level of detection).

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival time is defined as the time from randomization to death due to any cause. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: From registration to death due to any cause, assessed up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Bevacizumab and Nab-paclitaxel) | Arm B (Ipilimumab)
Number analyzed (Participants) | 12 | 12
months | 18.4 [11.4 to NA] — The 95% confidence interval upper limit was not reached (below the level of detection). | 27.0 [11.3 to NA] — The 95% confidence interval upper limit was not reached (below the level of detection).

3. Secondary Outcome: Number of Patients With Tumor Response
Description: Tumor response defined as complete or partial response using Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Complete response (CR): Disappearance of all evidence of disease, Partial response (PR): Regression of measurable disease and no new sites.
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Bevacizumab and Nab-paclitaxel) | Arm B (Ipilimumab)
Number analyzed (Participants) | 12 | 12
Participants
  CR | 2 | 0
  PR | 1 | 1

4. Secondary Outcome: The Number of Patients Who Experienced Toxicity
Description: The number of patients who experienced toxicity (grade 3 or higher adverse events considered at least possibly related to treatment) are reported below.
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Bevacizumab and Nab-paclitaxel) | Arm B (Ipilimumab)
Number analyzed (Participants) | 12 | 12
Participants | 9 | 7

5. Other Pre Specified Outcome: Changes in Biomarkers of Angiogenesis (Arm A)
Time Frame: Baseline to up to 5 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Changes in Biomarkers of Immunity
Time Frame: Baseline to up to 5 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Pharmacokinetic Changes in Paclitaxel Albumin-stabilized Nanoparticle Formulation Plasma Concentrations
Time Frame: Baseline, prior to the end of paclitaxel albumin-stabilized nanoparticle formulation infusion, and the morning after nab-paclitaxel infusion on days 1 and 8 of course 1
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 4 years
Description: Adverse events are reported for each arm group (i.e. Arm A, Arm B, Arm A Eligible for Crossover, and Arm B Eligible for Crossover)
Groups:
- Arm A Eligible for Crossover: Arm A patients who experienced progressive disease and eligible for crossover to Arm B AND evaluated for adverse events.
- Arm B Eligible for Crossover: Arm B patients who experienced progressive disease and eligible for crossover to Arm A AND evaluated for adverse events.
Arm/Group | Arm A (Bevacizumab and Nab-paclitaxel) | Arm B (Ipilimumab) | Arm A Eligible for Crossover | Arm B Eligible for Crossover
All-Cause Mortality (participants affected / at risk) | 10/12 | 8/12 | 6/7 | 5/7
Serious Adverse Events (participants affected / at risk) | 2/12 | 4/12 | 2/7 | 2/7
Other Adverse Events (participants affected / at risk) | 11/12 | 9/12 | 7/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Bevacizumab and Nab-paclitaxel) (N=12) | Arm B (Ipilimumab) (N=12) | Arm A Eligible for Crossover (N=7) | Arm B Eligible for Crossover (N=7)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Bevacizumab and Nab-paclitaxel) (N=12) | Arm B (Ipilimumab) (N=12) | Arm A Eligible for Crossover (N=7) | Arm B Eligible for Crossover (N=7)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 1 (3) | 1 (1) | 2 (2)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (5) | 2 (2) | 3 (7)
Diarrhea (Gastrointestinal disorders) | 2 (4) | 0 (0) | 2 (2) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Fatigue (General disorders) | 6 (7) | 2 (3) | 3 (3) | 6 (26)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papulopustular rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 9 (21) | 0 (0) | 1 (1) | 4 (11)
White blood cell decreased (Investigations) | 8 (19) | 0 (0) | 1 (1) | 3 (10)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 1 (1) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 1 (1) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (14) | 0 (0) | 1 (1) | 4 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 5 (9) | 2 (2) | 0 (0) | 2 (6)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-26): https://cdn.clinicaltrials.gov/large-docs/20/NCT02158520/Prot_SAP_000.pdf